CLINICAL TRIAL: NCT03737370
Title: A Phase I Trial of Fractionated Docetaxel and Radium 223 in Metastatic Castration-Resistant Prostate Cancer (CRPC)
Brief Title: Fractionated Docetaxel and Radium 223 in Metastatic Castration-Resistant Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: Bayer (Industry); Lahey Clinic (Other); Henry Ford Hospital (Other); Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IIR-US-2016-3279
Record Dates: First submitted 2018-10-25; First posted 2018-11-09 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Castrate Resistant Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; radium Ra 223 dichloride; Radium-223

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dose escalation (Experimental): There are four dose cohorts (1, 1a, 2, 2a) in this arm and two dose levels of docetaxel (40mg/m^2 [level 1] and 50mg/m^2 [level 2]). Dosing of Radium 223 remains the same in all cohorts (55 KBq/kg given every 28 days for 6 cycles).
  Maximum tolerated dose (MTD) of docetaxel will be assessed. MTD is defined as the highest dose-level, among those tested, associated with a rate of less than a 33% dose limiting toxicity (DLT).
  Interventions: Drug: Docetaxel; Radiation: Radium 223
- Dose expansion (Experimental): If the maximum tolerated dose (MTD) of docetaxel is found in arm 1, this dose level will be expanded to include an additional 25 subjects to confirm the safety and explore the preliminary anti-cancer effect. If the MTD is not identified, the study will be stopped and the expansion cohort will not be accrued.
  Interventions: Drug: Docetaxel; Radiation: Radium 223

INTERVENTIONS:
Drug: Docetaxel — Docetaxel will be administered every 2 weeks (on Day 1 and Day 15 of a 28 day cycle). Fractionated dosing dependent on cohort.
  Other Names: Fractionated Docetaxel
Radiation: Radium 223 — Radium 223 will be delivered every 28 days (on day 1) for 6 cycles.
  Other Names: Ra-223

SUMMARY:
The objective of this study is to determine the maximum safe dose of Ra-223 in combination with fractionated (split doses) docetaxel when given to subjects and to determine the best administering dose. The study will look at side effects that may happen while taking the combination treatment. A total of approximately 18 subjects will take part in the dose escalation part of the study and an additional 25 subjects will participate in the expansion cohort. This study will be conducted across four centers in the United States.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the safety and toxicity of a fractionated docetaxel schedule in combination with standard Ra-223.

Secondary Objectives include: assessment of progression-free survival, time to treatment failure, overall survival, ability of subjects to complete 6 cycles of the combination therapy, assessment of Prostate Specific Antigen (PSA) kinetics and objective responses (measurable disease), assessment of quality of life and assessment of bone bio-marker outcomes.

The study features a 4-week lead-in period with docetaxel monotherapy to assess for docetaxel intolerance. The lead-in period is then followed by combination therapy with Ra-223 every 4 weeks for 6 cycles in a traditional Phase I dose-escalation design.

A provision has been made to include prophylactic granulocyte colony stimulating factor (G-CSF) cohorts after the lead-in period if neutropenia is the dose limiting toxicity at either dose level.

The investigators hypothesize that the fractionated dosing of docetaxel will significantly mitigate the hematologic toxicity, preserve antineoplastic activity and allow for maintenance of the 4-weekly Ra-223 schedule.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed adenocarcinoma of the prostate
2. Documented metastatic castration resistant disease with PSA progression, radiographic progression, or both, despite medical or surgical castration
3. Two or more bone metastases detected on skeletal scintigraphy
4. Eligible for docetaxel chemotherapy
5. ECOG Performance Status 0-2
6. Adequate organ function:

   1. Hemoglobin > 10 g/dL
   2. Absolute Neutrophil Count ≥ 1,500 K/mL
   3. Platelet count ≥ 150,000 x 10^9/L
   4. Total bilirubin ≤ 1.5x upper limit of normal range, excluding Gilbert syndrome
   5. Serum AST ≤ 1.5 x upper limit of normal range
   6. Serum ALT ≤ 1.5 x upper limit of normal range
7. Estimated glomerular filtration rate (GFR) > 30mL/min
8. Ongoing castration (androgen deprivation therapy or prior orchiectomy)
9. Male subjects with female sexual partners of childbearing potential must agree to use at least one highly effective methods of birth control.
10. Ability to understand and willingness to sign an informed consent form prior to initiation of any study procedures.
11. Age ≥ 18 years

Exclusion Criteria:

1. Prior radionuclide therapy for CRPC
2. Prior docetaxel for CRPC. (Permitted if given for castration sensitive disease > 6 months prior).
3. Antiandrogen therapy within 4 weeks of enrollment. However, patients with primary failure of secondary anti-androgen therapy OR symptomatic progression, objective progression and/or biochemical evidence of rising PSA less than 4 weeks after discontinuation of anti-androgen therapy will not have anti-androgen withdrawal responses and will not be excluded.
4. Preexisting peripheral neuropathy grade 2 or higher.
5. Other serious medical condition as judged by the investigator.
6. Active second malignancy that requires therapy.
7. Known brain or leptomeningeal metastases
8. Concurrent enrollment in any other investigational anticancer therapy
9. Treatment with any myelosuppressive agent within 30 days of enrollment
10. Presence of bulky visceral metastases, defined as any of the following:

    1. ≥ 4 lung lesions (at least 1cm each in size in the longest diameter) or pulmonary lymphangitic metastasis
    2. Liver metastases with sum of lesion diameters totaling ≥ 5cm
11. Evidence of neuroendocrine or small cell differentiation on prior biopsy
12. History of severe hypersensitivity reactions to docetaxel or to drugs formulated with polysorbate 80

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLT) | Up to 29 Days
  DLT is defined as a subject in any cohort experiencing any of the following adverse events during cycle 1 of treatment, until cycle 2 day 1 of treatment: Thrombocytopenia (platelets < 75 x 10^9/L on C1D15 or < 100 x 10^9/L on C2D1), Neutropenia (ANC < 1000 K/mL on C1D15 or ANC < 1500 K/mL on C2D1), Grade 3 (by CTCAE v4) fatigue lasting ≥ 7 days, other non-hematologic toxicity ≥ grade 3, lasting ≥ 48 hours at least possibly related to treatment, or any toxicity (non-hematologic or hematologic) at least possibly related to treatment requiring dose reduction or dose interruption.

SECONDARY OUTCOMES:
Efficacy, assessed as non-progression/progression rate according to prostate cancer working group (PCWG2) criteria | From date of randomization until the date of first documented progression or death from any cause, whichever came first, assessed up to 25 years
  Time to progression of disease, calculated as a time-to-event endpoint
Progression Free Survival (PFS) | Up to 25 years
  Progression free survival is defined as the interval from first dose date of study drug to the earlier of the first documentation of definitive disease progression (assessed per PCWG2) or death from any cause
Time to Treatment Failure (TTTF) | Up to 25 years
  A measurement from the date of randomization to the first event which meets the criteria for disease progression (assessed per PCWG2 criteria) or death from any cause
Overall Survival | Up to 25 years
  Overall survival is defined as the interval from first dose date of study drug to death from any cause.
Proportion of Randomized Subjects to Complete Combination Therapy on Schedule per Protocol | Up to 28 weeks
  The number of subjects who were able to receive both lead-in doses of docetaxel and all 6 cycles of combination docetaxel and Ra223 on time (+/- 7 days).
Response to treatment, as assessed by prostate-specific antigen (PSA) Kinetics and Objective Responses | From date of randomization until the date of first documented progression or death from any cause, whichever came first, assessed up to 25 years
  Measurable disease calculated at each time point in which the data is collected. We will use mixed effect models to explore the temporal trajectories for the outcome changes over time in response to the treatment.
Satisfaction, as assessed by Quality of Life Questionnaires | From date of randomization until the date of first documented progression or death from any cause, whichever came first, assessed up to 25 years
  Measured by the Brief Pain Inventory (BPI) and Functional Assessment of Cancer Therapy (FACT-G) Questionnaires
Response to Treatment, as assessed by Bone Bio-marker Outcomes | Up to 28 weeks
  Measurement of bone-specific alkaline phosphatase and urine N-telopeptides (laboratory testing)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Mathew, MD, Principal Investigator — Tufts Medical Center
Locations (4):
- United States (4):
  - Lahey Hospital & Medical Center, Boston, Massachusetts
  - Tufts Medical Center, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parker C, Nilsson S, Heinrich D, Helle SI, O'Sullivan JM, Fossa SD, Chodacki A, Wiechno P, Logue J, Seke M, Widmark A, Johannessen DC, Hoskin P, Bottomley D, James ND, Solberg A, Syndikus I, Kliment J, Wedel S, Boehmer S, Dall'Oglio M, Franzen L, Coleman R, Vogelzang NJ, O'Bryan-Tear CG, Staudacher K, Garcia-Vargas J, Shan M, Bruland OS, Sartor O; ALSYMPCA Investigators. Alpha emitter radium-223 and survival in metastatic prostate cancer. N Engl J Med. 2013 Jul 18;369(3):213-23. doi: 10.1056/NEJMoa1213755. PMID 23863050
- [Background] Antonarakis ES, Lu C, Wang H, Luber B, Nakazawa M, Roeser JC, Chen Y, Mohammad TA, Chen Y, Fedor HL, Lotan TL, Zheng Q, De Marzo AM, Isaacs JT, Isaacs WB, Nadal R, Paller CJ, Denmeade SR, Carducci MA, Eisenberger MA, Luo J. AR-V7 and resistance to enzalutamide and abiraterone in prostate cancer. N Engl J Med. 2014 Sep 11;371(11):1028-38. doi: 10.1056/NEJMoa1315815. Epub 2014 Sep 3. PMID 25184630
- [Background] Antonarakis ES, Lu C, Luber B, Wang H, Chen Y, Nakazawa M, Nadal R, Paller CJ, Denmeade SR, Carducci MA, Eisenberger MA, Luo J. Androgen Receptor Splice Variant 7 and Efficacy of Taxane Chemotherapy in Patients With Metastatic Castration-Resistant Prostate Cancer. JAMA Oncol. 2015 Aug;1(5):582-91. doi: 10.1001/jamaoncol.2015.1341. PMID 26181238
- [Background] Oudard S, Banu E, Beuzeboc P, Voog E, Dourthe LM, Hardy-Bessard AC, Linassier C, Scotte F, Banu A, Coscas Y, Guinet F, Poupon MF, Andrieu JM. Multicenter randomized phase II study of two schedules of docetaxel, estramustine, and prednisone versus mitoxantrone plus prednisone in patients with metastatic hormone-refractory prostate cancer. J Clin Oncol. 2005 May 20;23(15):3343-51. doi: 10.1200/JCO.2005.12.187. Epub 2005 Feb 28. PMID 15738542
- [Background] Kellokumpu-Lehtinen PL, Harmenberg U, Joensuu T, McDermott R, Hervonen P, Ginman C, Luukkaa M, Nyandoto P, Hemminki A, Nilsson S, McCaffrey J, Asola R, Turpeenniemi-Hujanen T, Laestadius F, Tasmuth T, Sandberg K, Keane M, Lehtinen I, Luukkaala T, Joensuu H; PROSTY study group. 2-Weekly versus 3-weekly docetaxel to treat castration-resistant advanced prostate cancer: a randomised, phase 3 trial. Lancet Oncol. 2013 Feb;14(2):117-24. doi: 10.1016/S1470-2045(12)70537-5. Epub 2013 Jan 4. PMID 23294853
- [Background] Kantoff PW, Higano CS, Shore ND, Berger ER, Small EJ, Penson DF, Redfern CH, Ferrari AC, Dreicer R, Sims RB, Xu Y, Frohlich MW, Schellhammer PF; IMPACT Study Investigators. Sipuleucel-T immunotherapy for castration-resistant prostate cancer. N Engl J Med. 2010 Jul 29;363(5):411-22. doi: 10.1056/NEJMoa1001294. PMID 20818862
- [Background] Ryan CJ, Smith MR, de Bono JS, Molina A, Logothetis CJ, de Souza P, Fizazi K, Mainwaring P, Piulats JM, Ng S, Carles J, Mulders PF, Basch E, Small EJ, Saad F, Schrijvers D, Van Poppel H, Mukherjee SD, Suttmann H, Gerritsen WR, Flaig TW, George DJ, Yu EY, Efstathiou E, Pantuck A, Winquist E, Higano CS, Taplin ME, Park Y, Kheoh T, Griffin T, Scher HI, Rathkopf DE; COU-AA-302 Investigators. Abiraterone in metastatic prostate cancer without previous chemotherapy. N Engl J Med. 2013 Jan 10;368(2):138-48. doi: 10.1056/NEJMoa1209096. Epub 2012 Dec 10. PMID 23228172
- [Background] Beer TM, Armstrong AJ, Rathkopf DE, Loriot Y, Sternberg CN, Higano CS, Iversen P, Bhattacharya S, Carles J, Chowdhury S, Davis ID, de Bono JS, Evans CP, Fizazi K, Joshua AM, Kim CS, Kimura G, Mainwaring P, Mansbach H, Miller K, Noonberg SB, Perabo F, Phung D, Saad F, Scher HI, Taplin ME, Venner PM, Tombal B; PREVAIL Investigators. Enzalutamide in metastatic prostate cancer before chemotherapy. N Engl J Med. 2014 Jul 31;371(5):424-33. doi: 10.1056/NEJMoa1405095. Epub 2014 Jun 1. PMID 24881730
- [Background] Scher HI, Halabi S, Tannock I, Morris M, Sternberg CN, Carducci MA, Eisenberger MA, Higano C, Bubley GJ, Dreicer R, Petrylak D, Kantoff P, Basch E, Kelly WK, Figg WD, Small EJ, Beer TM, Wilding G, Martin A, Hussain M; Prostate Cancer Clinical Trials Working Group. Design and end points of clinical trials for patients with progressive prostate cancer and castrate levels of testosterone: recommendations of the Prostate Cancer Clinical Trials Working Group. J Clin Oncol. 2008 Mar 1;26(7):1148-59. doi: 10.1200/JCO.2007.12.4487. PMID 18309951
- [Background] Petrylak DP, Tangen CM, Hussain MH, Lara PN Jr, Jones JA, Taplin ME, Burch PA, Berry D, Moinpour C, Kohli M, Benson MC, Small EJ, Raghavan D, Crawford ED. Docetaxel and estramustine compared with mitoxantrone and prednisone for advanced refractory prostate cancer. N Engl J Med. 2004 Oct 7;351(15):1513-20. doi: 10.1056/NEJMoa041318. PMID 15470214
- [Background] Cessna JT, Zimmerman BE. Standardization of radium-223 by liquid scintillation counting. Appl Radiat Isot. 2010 Jul-Aug;68(7-8):1523-8. doi: 10.1016/j.apradiso.2009.11.068. Epub 2009 Dec 2. PMID 20097568
- [Background] Zimmerman BE, Bergeron DE, Cessna JT, Fitzgerald R, Pibida L. Revision of the NIST Standard for (223)Ra: New Measurements and Review of 2008 Data. J Res Natl Inst Stand Technol. 2015 Mar 11;120:37-57. doi: 10.6028/jres.120.004. eCollection 2015. PMID 26958437
- See also: Citation — http://ascopubs.org/doi/abs/10.1200/jco.2013.31.15_suppl.5021

DOCUMENTS (2):
  • Study Protocol (2018-10-02): https://cdn.clinicaltrials.gov/large-docs/70/NCT03737370/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-17): https://cdn.clinicaltrials.gov/large-docs/70/NCT03737370/SAP_001.pdf